CLINICAL TRIAL: NCT01148966
Title: A Phase 1 Study of Aminolevulinic Acid (ALA) to Enhance Visualization and Resection of Malignant Glial Tumors of the Brain
Brief Title: Aminolevulinic Acid During Surgery in Treating Patients With Malignant Brain Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7140; NCI-2010-00946 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2010-06-21; First posted 2010-06-23 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2013-05

CONDITIONS: Adult Anaplastic Astrocytoma; Adult Anaplastic Oligodendroglioma; Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma; Adult Mixed Glioma; Recurrent Adult Brain Tumor
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma; Glioblastoma; Gliosarcoma; Glioma; Brain Neoplasms | interventions — Aminolevulinic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (photodynamic therapy) (Experimental): Patients receive aminolevulinic acid PO 4 hours before undergoing surgery.
  Interventions: Drug: aminolevulinic acid; Other: laboratory biomarker analysis; Procedure: therapeutic conventional surgery

INTERVENTIONS:
Drug: aminolevulinic acid — Given PO
  Other Names: 5-ALA; 5-Aminolaevulinic Acid; ALA
Other: laboratory biomarker analysis — Correlative studies
Procedure: therapeutic conventional surgery — Standard brain tumor surgery with intra-operative frameless MRI stereotactic guidance and intra-operative ultrasound guidance

SUMMARY:
This phase I trial is studying the side effects and best dose of aminolevulinic acid during surgery in treating patients with malignant brain tumors. Aminolevulinic acid becomes active when it is exposed to a certain kind of light and may help doctors find and remove tumor cells during surgery

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES I. Establish a safe dose for oral ALA administration.

SECONDARY OBJECTIVES I. Determine which of 3 ALA (aminolevulinic acid) doses (10, 20 or 30 mg/kg) provide optimal discrimination between normal and malignant tissue intraoperatively.

II. Determine whether or not the use of ALA (compared to comparable cases performed without the aid of ALA) leads to a higher rate of gross total resection, as determined by postoperative MRI scanning within 48 hour of surgery completion.

III. Compare time-to-progression and survival to that in comparable cases performed without the aid of ALA.

OUTLINE: This is a phase I, dose-escalation study

Patients receive aminolevulinic acid orally (PO) 4 hours before undergoing surgery. After completion of study treatment, patients are followed up at week 5 and then every 8-12 weeks for 27 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients may have clinically documented primary malignant glioma for which re-resection is clinically indicated; in this instance, previous pathology slides will be reviewed by University of Washington Medical Center (UWMC) Neuropathology prior to surgery; alternatively, patients may have imaging studies (magnetic resonance imaging [MRI] and /or computed tomography [CT] scans), which are highly indicative of a new malignant glioma, for which surgical resection is clinically warranted; the anticipated histology at resection should include: glioblastoma, gliosarcoma, anaplastic astrocytoma, anaplastic oligodendroglioma, anaplastic oligoastrocytoma (mixed glioma)
* Prior therapy is not a consideration in protocol entry; patients with recurrence of known malignant gliomas are eligible following UWMC neuropathology slide review
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy is not a consideration for protocol entry
* Patients must have normal organ and marrow function as defined below:
* Leukocytes >= 3,000/uL
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 100,000/uL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 2.5 X institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* The effects of ALA on the developing human fetus are unknown; for this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Prior therapy is not an exclusion criterion
* Patients may not be receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ALA
* Personal or family history of porphyrias
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because ALA is of unknown teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ALA, breastfeeding should be discontinued if the mother is treated with ALA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-06; Primary Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Establishment of a safe dose for oral ALA administration | For 30 days post-aminolevulinic acid dose
  Using National Cancer Institute (NCI) Common Toxicity Criteria to quantify toxicity following ALA administration. We will use descriptive statistics to analyze the safety data, based on NCI toxicity criteria.
Determination of which of 3 ALA doses provide optimal discrimination between normal and malignant tissue intraoperatively | During surgery and from samples collected during surgery
  The results from three methods will be used collectively to determine whether or not it is prudent, safe and justified to proceed with 12 more patients using the highest dose tolerated without undue toxicity. The results from these three methods, both surgical fluorescence rating and neuropathologist ratings of fluorescence and presence, or absence, of tumor will be compared using a correlation coefficient.

SECONDARY OUTCOMES:
Comparison of time-to-progression (TTP) and survival to that in comparable cases performed without the aid of ALA | At week 5 and then every 8-12 weeks for 27 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Silbergeld, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States